CLINICAL TRIAL: NCT03676985
Title: An Open-label, Dose-escalation, Bi-weekly Phase I+II Clinical Trial in Treating Patients With Limited Stage of High-grade Osteosarcoma of Maintenance Therapy After Adjuvant Chemotherapy
Brief Title: A Clinical Study of PD-L1 Antibody ZKAB001(Drug Code) in Limited Stage of High-grade Osteosarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2017-03
Record Dates: First submitted 2018-09-13; First posted 2018-09-19 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZKAB001 5 mg/kg/time (Experimental): Three or six patients will treated with the dose of 5 mg/kg/time of ZKAB001 IV bi-weekly. DLT was observed within 28 days after administration.
  Interventions: Drug: ZKAB001 5mg/kg
- ZKAB001 10 mg/kg/time (Experimental): Three or six patients will treated with the dose of 10 mg/kg/time of ZKAB001 IV bi-weekly. DLT was observed within 28 days after administration.
  Interventions: Drug: ZKAB001 10mg/kg
- ZKAB001 15 mg/kg/time (Experimental): Three or six patients will treated with the dose of 15 mg/kg/time of ZKAB001 IV bi-weekly. DLT was observed within 28 days after administration.
  Interventions: Drug: ZKAB001 15mg/kg

INTERVENTIONS:
Drug: ZKAB001 5mg/kg — 5mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 5 mg/kg/time
Drug: ZKAB001 10mg/kg — 10mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 10 mg/kg/time
Drug: ZKAB001 15mg/kg — 15mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 15 mg/kg/time

SUMMARY:
This is a Phase 1+2, open-label, dose-escalation, and multidose study, aiming to investigate the safety, tolerability and pharmacokinetics of ZKAB001 (a fully human monoclonal antibody targeting the Programmed Death - Ligand 1 (PD-L1) membrane receptor on T lymphocytes and other cells of the immune system) administered every 14 days in subjects with limited stage of high-grade osteosarcoma of maintenance therapy after adjuvant chemotherapy.

DETAILED DESCRIPTION:
The study will consist of 4 periods: Screening (up to 28 days), Lead-in period (Day -28), Treatment (up to 24 cycles or 1 year, whichever occurs first), and Follow-up (up to 2 years). There will be a lead-in period on Day -28 for each dose escalation cohort in which the single-dose pharmacokinetics(PK) of ZKAB001 will be characterized prior to initiation of continuous dosing in the first cycle of treatment. The lead-in period duration, PK time-points, doses and/or regimens used in subsequent cohorts may be modified based on the exposure (AUC) observed during the lead-in period (although the number of PK samples will not be increased). Treatment of continuous dosing is up to 24 cycles or 1 year, until as per investigator's opinion, subjects experience disease progression (evaluated by RECIST 1.1), no clinical benefit, or intolerable toxicity. If investigators suspect subjects experience pseudoprogression or has evidence to prove "mixed response", subjects can continue to accept treatment as investigator decided.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily gives written informed consent to participate in the study.
2. Patients aged between 18 and 55 (inclusive).
3. To diagnosed with limited stage of high-grade osteosarcoma (AJCC stage I-III) by histologically, the patients must have received neoadjuvant chemotherapy and adjuvant chemotherapy and primary tumor radical surgery (R0). The end of adjuvant chemotherapy should less than 12 weeks. Chemotherapy regimens must contain doxorubicin (ADM)/epirubicin (EPI)/pirarubicin (THP)/doxorubicin liposome (PLD) and cisplatin (DDP), the minimum cumulative doses are ADM 360 mg/m2, EPI 450mg/m2, THP 300mg/m2, PLD 240 mg/m2 and DDP 480 mg/m2.
4. Eastern Cooperative Oncology Group（ECOG）performance status of 0 or 1, with estimated life expectancy of at least 3 months.
5. Adequate blood routine, hepatic and renal function:

1)neutrophil count (ANC) absolutely acuity≥1.5 x 109 / L; 2)platelet count≥80 x 109 / L; 3)hemoglobin≥90 g/L; 4)serum albumin≥28 g/L; 5)bilirubin≤1.5 x ULN（upper limit of normal）; 6)Alanine transaminase （ALT）and AST≤1.5 x ULN, serum Cr≤1.25 x ULN; 7) endogenous creatinine clearance≥50 ml/min (according Gault Cockcroft formula).

7.Female reproductive subjects should take effective contraception during the study period and within 3 months after the study treatment period. The serum or urine human chorionic gonadotropin（HCG） examination must be negative within 7 days before the subject is enrolled.

Exclusion Criteria:

1. Local recurrence or metastasis.
2. Any active autoimmune disease or history of autoimmune disease (such as, but not limited to, interstitial pneumonia, uveitis, enteritis, hepatitis, arthritis, nephritis, pituitary inflammation, hyperthyroidism, hypothyroidism, etc.); Patients with vitiligo or asthma in childhood, adult still need medical intervention; Patients need bronchodilators for medical intervention of asthma.
3. Patients are using immunosuppressive agents, or systemic, or absorbable topical corticosteroid medications to achieve immunosuppressive purposes (doses >10mg/day prednisone or equivalent), which is ongoing 2 weeks before enrollment.
4. Have received any form of organ transplantation, including allogeneic stem cell transplantation.
5. Known allergy to macromolecular protein inhibitors or any of the components of ZKAB001.
6. Suffering from other malignant tumors other than this diseases in 5 years except for skin basal cell and squamous cell carcinoma.
7. Central nervous system metastases with clinical symptoms (such as cerebral edema and brain metastases requiring corticosteroid intervention). Previous treatment with brain or meningeal metastasis, such as clinical stabilization (MRI) less than 2 months, or systemic corticosteroid (dose >10mg/day prednisone or equivalent) less than 2 weeks.
8. Patients with clinical symptoms or diseases of the heart that cannot be well controlled, such as heart failure above New York Heart Association（NYHA ）2 grade, unstable angina pectoris, myocardial infarction in 1 year, and clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, have left ventricular ejection fraction < 50% at rest in the ultrasound cardiogram.
9. Previous radiotherapy, chemotherapy, surgery or molecular targeted therapy, less than 3 weeks after treatment and before study drug; Patients whose adverse events caused by previous treatment did not recover to level 1 of CTCAE, except for hair loss.
10. Active infection, or unexplained fever> 38.5 degrees during screening period or before the first dose of ZKAB001 (subjects with fever from the tumor could be enrolled upon investigator's decision).
11. Human immunodeficiency virus (HIV) positive, syphilis spirochete positive, untreated active hepatitis.
12. The patient is participating in other clinical studies or is less than 1 month away from the end of the previous clinical study.
13. To receive other anti-tumor treatment during the study.
14. To treated with other PD-1 and/or PD-1, or CTLA-4（Cytotoxic T Lymphocyte Antigen-4）antibodies, or other drugs for immunomodulatory receptor preparations previously.
15. Recent history of prophylactic non-cancer vaccination (such as seasonal influenza vaccine and human papillomavirus（HPV）vaccine) within 28 days before screening.
16. History of mental drug abuse, alcohol abuse or drug abuse.
17. Pregnant or lactating women.
18. Any mental condition that prevents the understanding or provision of the informed consent.
19. It is determined by the investigator that the patient has other factors that may lead to the termination of the study, such as other serious diseases or serious laboratory test abnormalities or other factors that may affect the safety of the patients , family or social factors that may affect the study data and sample collection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2020-02-14 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days after first dose
  Adverse events of level 3 or above related to the study drug occurring within 28 days after the first dose as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Maximal tolerable dose(MTD) | 28 days after first dose
  DLT occurs in less than 1/6 subjects, this lower dose is defined as MTD.
EFS(event-free survival) | through study completion, an average of 3 years
  The rate of 3-year event-free survival
AUC(0-t) | 24 periods or 1 year
  Area under curve 0-t
AUC(INF) | 24 periods or 1 year
  Area under curve INF
Cmax | 24 periods or 1 year
  Peak concentration
Tmax | 24 periods or 1 year
  Peak time
T1/2 | 24 periods or 1 year
  Half life
Vss | 24 periods or 1 year
  Steady-state apparent volume of distribution based on plasma concentration
total body clearance（CLT） | 24 periods or 1 year
  total body clearance
Cmin | 24 periods or 1 year
  The trough value at steady state
the percentage of the receptors of PD-L1 in CD14+ monocytes and CD3+T cells | through study completion, an average of 3 years
  To detected the percentage of the receptors of PD-L1 in CD14+（cluster of differentiation 14+ ） monocytes and CD3+（cluster of differentiation 3+）T cells.
the number of subjects presenting detectable anti drug antibodies (ADAs) | through study completion, an average of 3 years
  To evaluated the number of subjects presenting detectable anti drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: yang Yao, master, Study Director — 600 yishan road, Shanghai
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903